CLINICAL TRIAL: NCT06109558
Title: A Prospective Clinical Research of Efficacy and Safety of LMV-12(HE003) Combined With Osimertini in the Treatment of Advanced Non-small Cell Lung Cancer That Has Previously Failed From EGFR Inhibitor Therapy
Brief Title: The Efficacy and Safety of LMV-12 Combined With Osimertinib in NSCLC
Acronym: PROFILE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Director of Clinical Trial, Hunan Province Tumor Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023049
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Non Small Cell Lung Cancer; RET Gene Mutation; MET Amplification; EGF-R Positive Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Patients with MET amplication（by FISH, NGS or IHC）
  Interventions: Drug: LMV-12(HE003)
- Cohort B (Experimental): Patients with RET fusion.
  Interventions: Drug: LMV-12(HE003)

INTERVENTIONS:
Drug: LMV-12(HE003) — 1 cycle was 28 days. LMV-12(HE003), 30mg or 60mg, continuously for 21 days, and the drug was discontinued for 7 days. Osimertinib, 80mg, continuously for 28 days.
  Other Names: Osimertinib

SUMMARY:
This is an open-label, single-arm, dose-escalation, multicenter phase I/II clinical trial. The primary endpoints of this study were to evaluated the safety, tolerability, pharmacokinetic profile and preliminary efficacy of HE003 in combination with osimertinib in patients with advanced solid tumors who have failed previous standard therapy. The secondary endpoints of this study were to evaluated the efficacy HE003 in combination with osimertinib in patients with advanced solid tumors who have failed previous standard therapy.

DETAILED DESCRIPTION:
This is an open-label, single-arm, dose-escalation, multicenter phase I/II clinical trial. The primary endpoints of this study were to evaluated the safety, tolerability, pharmacokinetic profile and preliminary efficacy of HE003 in combination with osimertinib in patients with advanced solid tumors who have failed previous standard therapy. The secondary endpoints of this study were to evaluated the efficacy HE003 in combination with osimertinib in patients with advanced solid tumors who have failed previous standard therapy.

The study were devided in several cohorts following the different subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects selected for this study must meet all of the following criteria:

  1. Sign written informed consent before implementing any trial-related procedures;
  2. Age ≥18 years old;
  3. No limit on the gender;
  4. Histological or cytological confirmed advanced or metastatic non-small cell lung cancer, ineligible for radical surgery, relapse after failure of previous treatment with first-line (including first, second, and third generation)EGFR inhibitors.

     Cohort A：MET amplification,(by FISH, NGS or IHC) Cohort B：RET fusion.
  5. Laboratory tests for organ function levels must meet the following requirements:

     1. Absolute neutrophil count ≥ 1.5 × 109/L;
     2. Platelet count ≥ 100 × 109/L;
     3. Hemoglobin ≥ 9 g/dL;
     4. Bilirubin ≤1.5 times ULN; e) AST and ALT ≤2.5 times ULN (total bilirubin ≤3 times the upper limit of normal and AST and ALT ≤5 times the upper limit of normal are permitted if hepatic metastases are present);

     f) Serum creatinine ≤ 1.5 times ULN or creatinine clearance ≥ 60 mL/min (according to the Cockcroft-Gault formula);
  6. For premenopausal women of childbearing potential a pregnancy test must be performed within 7 days prior to initiation of treatment, a serum pregnancy test must be negative, and they must be non-lactating; all enrolled patients (whether male or female) should use adequate barrier contraception throughout the treatment period and for 3 months after completion of treatment.

Exclusion Criteria:

1. Subjects treated with CYP isozyme inducers or inhibitors (see Appendix 4 for details) within 3 weeks prior to enrollment;
2. Pregnant or lactating women;
3. History of immunodeficiency or other acquired, congenital immunodeficiency diseases;
4. Patients with prior bone marrow transplantation or prior solid organ transplantation;
5. Patients with a combination of gastrointestinal perforation, gastrointestinal fistula, or non-gastrointestinal fistula;
6. Prior history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy, or any evidence of clinically active interstitial lung disease.
7. Hepatitis B, hepatitis C, or human immunodeficiency virus (HIV-positive). Hepatitis B is eligible for this study at <500 IU/mL (or 2500 cps/mL) by quantitative HBV-DNA testing, and hepatitis C (HCV) antibody-positive patients are eligible for this study only if the polymerase chain reaction shows HCV RNA negativity;
8. Fulfillment of any of the following cardiac criteria: (i) Bazetts' mean corrected QT interval (QTc) derived from electrocardiogram (ECG) examination at rest >470 msec (women) or >450 msec (men) (in the case of the 1st abnormality, retested once within 48 h and calculated by averaging the results of the 2 times); and (ii) a wide variety of clinically significant rhythmic, conduction, and resting ECG morphologic Abnormalities, such as complete left bundle branch block, grade III conduction block, grade II conduction block, PR interval >250 msec; (iii) Myocardial ischemia or myocardial infarction of grade I or higher, or congestive heart failure of grade ≥2 (New York Heart Association (NYHA) classification); (iv) Factors that may increase the risk of prolongation of QTc or the risk of arrhythmic events, such as coronary artery disease, heart failure hypokalemia, congenital long QT syndrome, family history of a first-degree relative with long QT syndrome or sudden unexplained death before the age of 40, and ongoing use of any medication known to prolong the QT interval;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-31 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
ORR | Time from first subject dose to study completion, or up to 36 month
  Defined as the proportion of subjects in complete remission (CR) and partial remission (PR) to the total subjects
Adverse event and safety | Time from first subject dose to study completion, or up to 36 month
  Number of participants experiencing clinical and laboratory adverse events (AEs)

SECONDARY OUTCOMES:
PFS | Time from first subject dose to study completion, or up to 36 month
  Progression free survivaltime, define as first dose to the disease progression death of the subject due to any cause
OS | Time from first subject dose to study completion, or up to 36 month
  Overral survival time, define as first dose to the death of the subject due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Nong Yang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China